CLINICAL TRIAL: NCT06502483
Title: Treatment Development Study of the Promoting Resilience in Stress Management (PRISM) Intervention for Depression and Anxiety in Young Adults With Cancer
Brief Title: PRISM for Depression and Anxiety in Young Adults With Cancer
Acronym: PRISM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Samantha Bento, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-147
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer Diagnosis; Non-Metastatic Neoplasm; Anxiety; Anxiety Disorders; Depression; Depressive Disorder; Depression, Anxiety; Desmoid
Keywords: Cancer Diagnosis; Non-Metastatic Neoplasm; Anxiety; Anxiety Disorders; Depression; Depression Disorder; Depression, Anxiety; Young adults with cancer; Desmoid tumor
MeSH Terms: conditions — Anxiety Disorders; Depression; Depressive Disorder; Desmoid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRISM Program (Experimental): Participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with questionnaires.
  * 6 weekly or bi-weekly remote or in-clinic, psychotherapy sessions with psychologist.
  * Final questionnaires and post-study exit interview
  Interventions: Behavioral: Promoting Resilience in Stress Management Program

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management Program — Promoting Resilience in Stress Management (PRISM; Rosenberg et al., 2018; Rosenberg et al., 2021) is is an evidence-based skills-based resilience intervention. In the current study, PRISM sessions with be facilitated by a trained mental health provider to equip participants with skills for coping with anxiety, low mood, and adjustment to cancer diagnosis and to target four resilience resources (i.e., stress management, goal setting, cognitive reframing, and meaning-making). Sessions will be conducted by phone or Zoom, a HIPAA-compliant telemedicine platform. The optional mPRISM phone application includes 6 modules to practice PRISM skills and is available for iOS/Android.
  Other Names: PRISM Program

SUMMARY:
This research study is being done to test the feasibility of an existing supportive program (PRISM) to address psychological symptoms (i.e., depressive and anxiety symptoms) that young adult participants diagnosed with cancer or desmoid tumor may experience.

The name of the intervention used in this research study is:

-Promoting Resilience in Stress Management (PRISM) Program

DETAILED DESCRIPTION:
This research study is being done to test the initial feasibility and acceptability of a six-session, skills-based resilience coaching intervention, Promoting Resilience in Stress Management (PRISM; Rosenberg et al., 2018; Rosenberg et al., 2021), that targets four resilience resources (stress management, goal setting, cognitive reframing, and meaning-making) for young adult patients (18-30 years old) with cancer or desmoid tumor who are treated with curative intent and who report moderate depressive and/or anxiety symptoms.

The research study procedures include screening for eligibility, completing one diagnostic assessment of depressive and anxiety symptoms, pre-intervention and post-intervention questionnaires, completion of the six-session PRISM intervention, and a semi-structured exit interview about the experience with the PRISM intervention.

Participation in this research study is expected to last approximately 2 to 3 months.

It is expected that up to 15 young adults with cancer (i.e., participants) and up to a total of 15 support persons (i.e., friends or family members who participants will have an option to invite for the final session of the intervention) will take part in this research study.

The Hans and Mavis Lopater Foundation is funding this research study by providing philanthropic support.

ELIGIBILITY:
Inclusion Criteria for Participants:

1. 18-39 years of age
2. Speak and comprehend English sufficiently to be able to complete study procedures and participate in the program in English*
3. Have been diagnosed with cancer or desmoid tumor at least 6 or more weeks ago
4. Currently receiving treatment or has completed treatment for cancer or desmoid tumor no more than 6 months ago
5. Score 10-24 (with question #9 not endorsed, or 0) on the PHQ-9 (Kroenke et al., 1999) or/and score 10-21 on the GAD-7 (Spitzer et al., 2006) during the initial screening assessment.

Participant Exclusion Criteria:

1. Adults unable to consent, individuals who are not yet adults (age <18), pregnant women, and prisoners.
2. Individuals who score less than 10 on both PHQ-9 and GAD-7.
3. Individuals who are diagnosed with cancer less than 6 weeks at the time of screening (we will be able to approach them again after 6 weeks since diagnosis has passed), or those who completed treatment more than 6 months ago will also be ineligible for this study; they will be offered resources for support, if desired.

5) Individuals who report any suicidality (ideation, plan, and/or intent) on PHQ-9 screen (i.e., endorse anything more than 0 for question #9) at the time of the eligibility screening will also be excluded from the current study, and the appropriate safety measures and/or referral to a mental health provider will be made (see section 14.1 for more details on the procedure).

Inclusion Criteria for Support Person:

-≥ 18 years of age

-A friend or family member invited by the study participant to join the 6th PRISM session

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of PRISM Intervention Completion | Up to 12 weeks
  Feasibility is defined as 70% of PRISM sessions are completed by participants who start the study.
Rate of Study Assessment Completion | Up to 12 weeks
  Study feasibility is defined as 70% of all study assessments are completed by participants who complete PRISM sessions.
Participant Satisfaction | At final intervention session, up to 6 weeks
  Acceptability of the PRISM intervention will be determined by responses on semi-structured exit interviews using descriptive statistics and scores on the Client Satisfaction Questionnaire- (CSQ-8), an 8-item measuring a participant's opinions and assessment of the intervention. Total scores range from 8 to 32 with a higher number indicating greater satisfaction.

SECONDARY OUTCOMES:
mPRISM Phone Application Usage | Up to 12 weeks
  The feasibility of the mPRISM phone application as a tool to practice PRISM skills, as evidenced by the participant usage metrics.
Questionnaires | Up to 12 weeks
  The feasibility of using the assessment questionnaires in the current study (e.g., length, administration)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Bento, PhD, Principal Investigator — Dana-Farber Cancer Institute; Greta J Khanna, PhD, MA, Study Director — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Background] Rosenberg AR, Bradford MC, McCauley E, Curtis JR, Wolfe J, Baker KS, Yi-Frazier JP. Promoting resilience in adolescents and young adults with cancer: Results from the PRISM randomized controlled trial. Cancer. 2018 Oct 1;124(19):3909-3917. doi: 10.1002/cncr.31666. Epub 2018 Sep 19. PMID 30230531
- [Background] Rosenberg AR, Zhou C, Bradford MC, Salsman JM, Sexton K, O'Daffer A, Yi-Frazier JP. Assessment of the Promoting Resilience in Stress Management Intervention for Adolescent and Young Adult Survivors of Cancer at 2 Years: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2136039. doi: 10.1001/jamanetworkopen.2021.36039. PMID 34817581
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke, K., Spitzer, R. L., & Williams, J. B. W. (1999). Patient Health Questionnaire-9 (PHQ-9) [Database record]. APA PsycTests. https://doi.org/10.1037/t06165-000